CLINICAL TRIAL: NCT04708106
Title: A Randomized, Multi-Center, Open-Label, Parallel-Cohort Study to Characterize Product Use in Smokers Switching From Combustible Cigarettes to a RELX Electronic Nicotine Delivery System (ENDS)
Brief Title: Characterization of Product Use in Smokers Switching From Cigarettes to a RELX Electronic Nicotine Delivery System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cheerain HK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RELX-003
Record Dates: First submitted 2021-01-08; First posted 2021-01-13 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Electronic Cigarette Use
Keywords: Electronic Nicotine Delivery System; Biomarkers; Subjective Effects; Topography; E-cigarette
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RELX ENDS Tobacco Flavor (Experimental): Switch from combustible cigarettes to RELX ENDS Tobacco Flavor for 56 days
  Interventions: Other: RELX ENDS Tobacco Flavor
- RELX ENDS Menthol Flavor (Experimental): Switch from combustible cigarettes to RELX ENDS Menthol Flavor for 56 days
  Interventions: Other: RELX ENDS Menthol Flavor
- RELX ENDS Tobacco and Menthol Flavors (Experimental): Switch from combustible cigarettes to RELX ENDS Tobacco and Menthol Flavor for 56 days
  Interventions: Other: RELX ENDS Tobacco and Menthol Flavors
- Continue-smoking (No Intervention): Continue smoking combustible cigarettes for 56 days

INTERVENTIONS:
Other: RELX ENDS Tobacco Flavor — Ad libitum use of the RELX ENDS Tobacco Flavor product
  Arms: RELX ENDS Tobacco Flavor
Other: RELX ENDS Menthol Flavor — Ad libitum use of the RELX ENDS Menthol product
  Arms: RELX ENDS Menthol Flavor
Other: RELX ENDS Tobacco and Menthol Flavors — Ad libitum use of the RELX ENDS Tobacco and Menthol Flavor products
  Arms: RELX ENDS Tobacco and Menthol Flavors

SUMMARY:
The study will assess product use behaviors, biomarkers of exposure, subjective effects, and safety in smokers who switch to a RELX ENDS over 8-weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provides voluntary consent to participate in the study as documented on the signed informed consent form (ICF).
2. Is 22 to 65 years of age, inclusive, at the time of consent.
3. Is willing to comply with the requirements of the study.
4. Reports typically smoking 5 or more combustible CPD at Screening.
5. Has been a daily smoker for at least 12 months prior to Screening. Brief periods of non-smoking (e.g., up to ~7 consecutive days due to illness, trying to quit, participation in a study where smoking was prohibited) ≥ 56 days prior to Screening will be permitted at the discretion of the Investigator.
6. Has a positive urine cotinine test (≥ 200 ng/mL) at Screening and Test Visit 1.
7. Has an exhaled carbon monoxide (ECO) value > 10 ppm at Screening and Test Visit 1.
8. Has daily access to a cell phone for daily product use reporting.
9. If female, meets one of the following criteria:

If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 30 days prior to the first product use and during the study. An acceptable method of contraception includes one of the following:

* Abstinence from heterosexual intercourse
* Hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
* Intrauterine device (with or without hormones) OR agrees to use a double barrier method (e.g. condom and spermicide) during the study.

If a female of non-childbearing potential - should be surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (at least 1 year without menses), as confirmed by follicle stimulating hormone (FSH) levels.

Exclusion Criteria:

1. Has a history or presence of clinically significant uncontrolled gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. Has a clinically significant abnormal finding on the physical examination, medical history, vital signs, electrocardiogram (ECG), or clinical laboratory results, in the opinion of the Investigator.
3. Has a positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at Screening.
4. Has a positive COVID-19 test at Screening or during the study.
5. Has had an acute illness (e.g., upper respiratory infection, viral infection) within 14 days prior to Test Visit 1.
6. Has a fever (> 100.5°F) at Screening or Test Visit 1.
7. Has a body mass index (BMI) greater than 40.0 kg/m2 or less than 18.0 kg/m2 at Screening.
8. Has a systolic blood pressure < 90 mmHg or > 150 mmHg, diastolic blood pressure < 40 mmHg or > 95 mmHg, or heart rate < 40 bpm or > 99 bpm at Screening.
9. Has a post-bronchodilator forced expiratory volume in 1 second:forced vital capacity (FEV1:FVC) ratio < 0.7 and FEV1 < 50% of predicted at Screening.
10. Has a post-bronchodilator FEV1 increase ≥ 12% and > 200 mL from pre- to post-bronchodilator at Screening.
11. Has used an ENDS product on >7 days during each of the 3 months prior to Screening or any use from Screening to Test Visit 1 other than as may be required for this study.
12. Reports use of a very-low nicotine content cigarette (e.g., Moonlight, Spectrum, VLN) as usual brand.
13. Has used nicotine-containing products other than manufactured cigarettes (e.g., ENDS products (e-cigarettes), roll-your-own cigarettes, bidis, snuff, nicotine inhaler, pipe, cigar, chewing tobacco, nicotine patch, nicotine spray, nicotine lozenge, or nicotine gum) within 14 days prior to Test Visit 1.
14. Has used any products for the purpose of smoking cessation, including, but not limited to, nicotine replacement therapies, varenicline (Chantix), or buproprion (Zyban) from 30 days prior to Screening through the duration of the study.
15. Is a self-reported puffer (i.e., draws smoke from the cigarette into the mouth and throat but does not inhale).
16. Is postponing a planned smoking quit attempt in order to participate in the study.
17. Has a history of drug or alcohol abuse within 12 months prior to Screening, as determined by the Investigator.
18. Is allergic to PG or glycerin.
19. Has a positive urine drug or alcohol breath test at Screening or Test Visit 1. At the discretion of the investigator, a subject testing positive for tetrahydrocannabinol may be permitted to participate if the subject reports use by routes other than inhalation.
20. If female, the subject is pregnant, breastfeeding, or intends to become pregnant from Screening through the duration of the study.
21. Has been treated for depression, diabetes, asthma, emphysema, or chronic obstructive pulmonary disease within 12 months prior to Test Visit 1.
22. Has previously been diagnosed with any form of cancer, except for basal cell or squamous epithelial carcinomas of the skin that have been resected at least 12 months prior to Screening 1.
23. Has a planned surgery that would occur during study participation.
24. Has participated in a previous clinical study for an investigational drug, device, biologic, or tobacco product within 30 days prior to Test Visit 1.
25. Is or has a first-degree relative (e.g., spouse, parent, sibling, or child) who is a current or former employee of a tobacco or ENDS manufacturer or is a named party or class representative in litigation with the tobacco or ENDS industry.
26. Is or has a first-degree relative (e.g., spouse, parent, sibling, or child) who is a current employee of the clinic site.
27. Is or has a first-degree relative (e.g., spouse, parent, sibling, or child) who is a current employee of the Sponsor.
28. Has previously taken part in (from completion of any baseline measurements), has been withdrawn from, or has completed this study.
29. In the opinion of the Investigator, the subject should not participate in this study.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Weekly RELX ENDS product use | 56 days
  Self-reported number of RELX ENDS pods started each week.
Daily number of cigarettes smoked | 56 days
  Self-reported number of cigarettes smoked daily by study week.
Number of puffs from the RELX ENDS each day | 56 days
  Self-reported number of puffs from the RELX ENDS daily by study week (0, < 100, ≥ 100 per day).

SECONDARY OUTCOMES:
Biomarkers of exposure measured in blood | Baseline, Day 28, and Day 56
  Change in carbon monoxide concentration in the blood.
Biomarkers of tobacco exposure measured in urine | Baseline, Day 28, and Day 56
  Change in creatinine-adjusted NNAL, NNN, 3-HPMA, CEMA, HMPMA, S-PMA, HEMA, 1-OHP, o-toluidine, nicotine equivalents, and propylene glycol excreted in urine.
Subjective effects as measured by the Penn State [Electronic] Cigarette Dependence Index (PS[E]CDI) | Baseline, Day 14, Day 28, Day 42, and Day 56
  Change in product dependence as measured by the PSCDI/PSECDI total score. Total scores may range for 0 to 20, with higher levels of dependence associated with higher scores.
Subjective effects as measured by the Cough Questionnaire | Baseline, Day 14, Day 28, Day 42, and Day 56
  Change in self-reported cough symptoms as measured by responses to the Cough Questionnaire.
Subjective effects as measured by the Questionnaire of Smoking Urges-Brief (QSU-Brief) | Baseline, Day 14, Day 28, Day 42, and Day 56
  Change in smoking urge as measured by the QSU-Brief factor 1 and factor 2 scores. Questionnaire responses are measured on a Likert scale range of 1 [not at all] to 7 [extremely].
Subjective effects as measured by the Minnesota Tobacco Withdrawal Scale-Revised (MTWS-R) | Baseline, Day 14, Day 28, Day 42, and Day 56
  Change in withdrawal symptoms as measured by the MTWS-R total score, which includes the DSM-5 and craving items from the Minnesota Tobacco Withdrawal Scale. Questionnaire responses are measured on a Likert scale range of 0 [none] to 4 [severe]).
Subjective effects as measured by the Modified Product Evaluation Scale (mPES) | Baseline, Day 14, Day 28, Day 42, and Day 56
  Change in product assessments as measured by mPES satisfaction, psychological reward, aversion, and relief subscale scores. Questionnaire responses are measured on a Likert scale range of 1 [not at all] to 7 [extremely].
Subjective effects as measured by the Future Intent to Use Questionnaire | Baseline, Day 14, Day 28, Day 42, and Day 56
  Change in future intent to use cigarettes and ENDS products as measured by responses to the Future Intent to Use Questionnaire. Questionnaire responses are measured on a Likert scale range of 1 [extremely unlikely] to 7 [extremely likely].
Subjective Effects as measured by the Health Effects Perceptions Questionnaire | Baseline and Day 56
  Harmful and addictiveness perceptions as measured by responses to the Health Effects Perceptions Questionnaire.
Puff topography - number of puffs | Baseline, Day 28, and Day 56
  Change in the number of puffs during a 1-hour puff topography session.
Puff topography - puff duration | Baseline, Day 28, and Day 56
  Change in puff duration during a 1-hour puff topography session.
Puff topography - puff volume | Baseline, Day 28, and Day 56
  Change in puff volume during a 1-hour puff topography session.
Puff topography - peak puff flow rate | Baseline, Day 28, and Day 56
  Change in peak puff flow rate during a 1-hour puff topography session.
Puff topography - average flow rate | Baseline, Day 28, and Day 56
  Change in average flow rate during a 1-hour puff topography session.
Puff topography - inter-puff interval | Baseline, Day 28, and Day 56
  Change in inter-puff interval during a 1-hour puff topography session.
RELX ENDS product use | Day 28 and Day 56
  Change in pod weight during a 1-hour topography session
Incidence of product-use emergent adverse events [Safety and Tolerability] | 56 days
  Incidence of product-use emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Donald Graff, PharmD, Study Director — Sponsor Representative; Mark Adams, MD, Principal Investigator — AMR - Lexington
Locations (5):
- United States (5):
  - Pillar Clinical Research, Bentonville, Arkansas
  - AMR - Lexington, Lexington, Kentucky
  - QPS, Springfield, Missouri
  - AMR - Las Vegas, Las Vegas, Nevada
  - AMR - Knoxville, Knoxville, Tennessee